CLINICAL TRIAL: NCT01772745
Title: The Comparison of Single Incision Laparoscopic Cholecystectomy and Three Port Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, manuk norayk manukyan, Ass.Prof., Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mütf3
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Gallbladder Disease
Keywords: single incision; cholecystectomy; laparoscopy
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): SILS cholecystectomy
  Interventions: Procedure: SILS cholecystectomy
- Group 2 (Active Comparator): TPCL cholecystectomy
  Interventions: Procedure: TPCL cholecystectomy

INTERVENTIONS:
Procedure: SILS cholecystectomy — Single incision laparoscopic cholecystectomy will be performed
  Arms: Group 1
Procedure: TPCL cholecystectomy — Three port laparoscopic cholecystectomy will br performed
  Arms: Group 2

SUMMARY:
Laparoscopic techniques have allowed surgeons to perform complicated intrabdominal surgery with minimal trauma. Laparoscopic cholecystectomy has been recognized since 1987 as the gold standard procedure for gallbladder surgery. Single incision laparoscopic surgery (SILS) was developed with the aim of reducing the invasiveness of conventional laparoscopy. In this study we aimed to compare results of SILS cholecystectomy and three port conventional laparoscopic (TPCL) cholecystectomy prospectively

DETAILED DESCRIPTION:
Single-incision laparoscopic procedures have evolved gradually to include a multitude of various surgeries. The current literature documents the use of a single-incision or single-port access surgery for cholecystectomies, adrenalectomies, splenectomies, appendectomies, herniorrhaphies, bariatrics, and colon surgery.

Total of 100 patients who undergoing laparoscopic cholecystectomy for gallbladder disorders will randomly assign to undergo SILS cholecystectomy group (n = 50) or TPCL cholecystectomy group (n= 50) according to a computer-generated table of random numbers. Demographics (ie, age, gender, body mass index (BMI), American Society of Anesthesiology (ASA) score, indication for operation, need for conversion to a standard or three port laparoscopic cholecystectomy, need for conversion to an open cholecystectomy will be recorded. Outcome measures include operative morbidity, operative time, pain score, hospital stay. Morbidity will be evaluated by rates of bile leak, wound infection, hospital readmission, and hernia.

ELIGIBILITY:
Inclusion Criteria:

* Required laparoscopic cholecystectomy for gallbladder disease.

Exclusion Criteria:

* American Society of Anesthesiologists score (ASA) more than III,
* Patients had prior abdominal surgery,
* Patients admitted outside working hours with acute cholecystitis,
* Patients have choledocolithiasis,
* pregnancy,
* ongoing peritoneal dialysis,
* lack of written informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
pain score | Postoperative first 24 hours
  Postoperative pain will be assessed according Visual analog scale from 0 (no pain) to 10 (worst pain imaginable. Postoperative six hour VAS (POSH-VAS) and postoperative first day VAS (POFD-VAS) will be recorded and compared.
Intraoperative complications | Average of 70 minutes
  Per operative complications will be recorded.
  * Bleeding
  * Gallbladder perforation
  * Bile leakage
  * Bowel perforation
  * Complications associated with increased intra-abdominal pressure

SECONDARY OUTCOMES:
Operating time | Average of 70 minutes
  The operating time will be defined as the time from the first incision to the last suture's placement.

OTHER OUTCOMES:
Length of hospital stay | Average of 2 days
  Length of hospital stay will be recorded postoperative period.
Postoperative complications | 24th hour, 2nd day, 3rd day, 7th day, 1st month, 3rd month, 6th month, 1st year
  Postoperative complications will be recorded postoperative follow up.
  * Bleeding
  * Bile leakage
  * Intrabdominal injury
  * Wound infection
  * Port site hernia

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Deveci, Ass. Prof., Principal Investigator — Maltepe University, School of Medicine , General Surgery Department; Manuk N. Manukyan, Ass.Prof., Study Director — Maltepe University, School of Medicine, General Surgery Department; Umut Barbaros, Ass.Prof., Principal Investigator — Istanbul University, Istanbul Medical School, General Surgery Department; Abut Kebudi, Prof., Study Chair — Maltepe University, School of Medicine, General Surgery Department; Sertan Kapakli, Ass.Prof., Principal Investigator — Maltepe University, School of Medicine, General Surgery Department

REFERENCES:
- [Derived] Deveci U, Barbaros U, Kapakli MS, Manukyan MN, Simsek S, Kebudi A, Mercan S. The comparison of single incision laparoscopic cholecystectomy and three port laparoscopic cholecystectomy: prospective randomized study. J Korean Surg Soc. 2013 Dec;85(6):275-82. doi: 10.4174/jkss.2013.85.6.275. Epub 2013 Nov 26. PMID 24368985